CLINICAL TRIAL: NCT04292691
Title: Double-blinded Randomised Controlled Trial (RCT) Comparing a High Ankle Block to Placebo in Patients Treated for Ankle Pathologies
Brief Title: High Ankle Block in Ankle Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Sebastian. F. Baumbach, Principal investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-1
Record Dates: First submitted 2020-02-25; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Ankle Fractures; Anesthesia, Local
Keywords: Ankle fracture; Foot block; Perioperative pain management
MeSH Terms: conditions — Ankle Fractures | interventions — Ropivacaine; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Double blinded, randomised control trial
Who Masked: Participant, Care Provider
Masking Description: Randomization will be conducted by the Principle Investigator through RedCap. The syringe is prepared under sterile setting in a separate room by a nurse not involved in any further part of the medical treatment. The syringe with unknown content will be handed to the anaesthesiologist performing the anaesthesia. Therefore the anaesthesiologist performing the block as well as the guiding the anaesthesia throughout the surgery does not know what was injected.
  The total intraoperative morphine milligram equivalent dose will be automatically drawn from our anaesthesia recording program (NarcoData) and the cumulative morphine milligram equivalent dose use between skin incision and beginning Recovery Room calculated. The patient than receives the Piritramid PCA and the total morphine milligram equivalent dose use will again be drawn automatically from the machine. The VAS Score will be entered by the patient in a tablet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine (Experimental): A cumulative amount of approx. 40ml ropivacaine 0.5% (≙400mg (2x200mg) ropivacaine) is applied immediately before surgery. They are applied in a ring wall 10 cm cranially of the tip of the medial and lateral malleolus (N. peroneus superficialis (N. cutaneus dorsalis medius et intermedius, N. saphenus, N. suralis), as well as sonographically controlled (N. peroneus profundus and N. suralis)
  Interventions: Drug: 40ml of Ropivacaine 0.5% Injectable Solution
- Ringer's Lactate (Placebo Comparator): Analog to the Experimental Arm, but the same amount of Ringer (40ml) will be plicated instead Ropivacaine
  Interventions: Drug: 40ml of Ringer's Lactate

INTERVENTIONS:
Drug: 40ml of Ropivacaine 0.5% Injectable Solution — already outlined in the arm/group description
  Arms: Ropivacaine
Drug: 40ml of Ringer's Lactate — already outlined in the arm/group description
  Arms: Ringer's Lactate

SUMMARY:
The aim of the herein presented double-blinded is to compare the effectiveness of the high foot block against placebo infiltration in simple, uni- and bimalleolar ankle fractures.

Included will be all adult patients (>18a) treated surgically at our department. The standard peri-operative procedure at our clinic will no be altered but the additional high ankle block. The intraoperative opioid requirement, the Visual Analogue Scale for Pain (VAS) and the postoperative opioid requirement will be assessed and compared between the two groups

DETAILED DESCRIPTION:
Ankle fractures were among the most common injuries of the lower extremity. Peri-operative, multimodal pain therapy is of great importance in the surgical treatment of those injuries. Whereas simple (uni- and bimalleolar) ankle fractures are covered peri-operatively by oral pain medication and Piritramid-PCA (PCA=Patient-controlled analgesia), complex, trimalleolar fractures usually receive additional regional pain catheters (femoralis blockade and ischiadicus blockade).

Regional pain catheters have the major downside of motor paresis and are therefore critically discussed. Various studies have explored new techniques for perioperative pain therapy. An established procedure in midfoot and forefoot surgery is the foot block. It can be inserted at different heights around the ankle joint. However, the effectiveness of the high foot block has not yet been investigated for ankle fractures. The aim of the herein presented double-blinded is to compare the effectiveness of the high foot block against placebo infiltration in simple, uni- and bimalleolar ankle fractures.

All patients who are operated on in our department due to a uni- or bimalleolar ankle fracture, who are over 18 years of age and have no serious pre-existing conditions or contraindications to local anaesthesia (LA) are eligible for inclusion.

The perioperative procedure does not change to the current treatment standard at the University Hospital Munich - Ludwig Maximilians University (LMU) except for randomization for high foot block or placebo. Both the anesthesia and the postoperative pain therapy correspond to the current treatment standard and are the same for both groups. The intraoperative opioid requirement, the VAS and the postoperative opioid requirement will be assessed.

The data is collected using the RedCap database (#19-177), which has already been reviewed by the ethics committee. The evaluation will be performed using SPSS 25.0 (IBM).

ELIGIBILITY:
Inclusion Criteria:

* Age >17 years and <71 years
* Glomerular filtration rate (GFR) > 60
* American Society of Anaesthesiologists physical status classification system (ASA) < 4
* Independently mobile without aids before an accident
* Informed consent
* Uni- or bimalleolar (medial and lateral malleolus) ankle fractures requiring surgery

Exclusion Criteria:

* Age <18 years; >70 years
* GFR < 60
* ASA > 3
* Trimalleolar fractures or fractures necessitating open reduction and internal fixation (ORIF) of the posterior malleolus
* Not able to walk without aids (stick, rollator, etc.)
* Allergy to local anesthetics or drugs of the postOP pain regime
* Peripheral polyneuropathy
* Peripheral artery disease (PAD) grade IV°
* Dementia
* Depression, anxiety disorders or sleep disorders 18
* Pregnancy
* Denial of study participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative morphine milligram equivalent dose during the surgery (skin incision - recovery room) | Begin anaesthesia to begin recovery room; the time will vary between 1 and 4 hours
  The morphine equivalent doses will be calculated based on the morphines given throughout the surgery: Begin anaesthesia to begin recovery room
  Cumulative morphine milligram equivalent dose during the surgery (skin incision - recovery room)

SECONDARY OUTCOMES:
Visual Analogue pain Scale (VAS) | Will be collected at arrival at the recovery room and then 2 hours, 4 hours, 6 hours thereafter. For the further in-house duration,the VAS will be collected at 08:00 and 21:00 o'clock every day for further two days
  Postoperative pain measured on a 0-100 Visual Analogue pain Scale (VAS) with 0 meaning no pain and 100 most sever pain imaginable
Postoperative cumulative morphine milligram equivalent dose | The Piritramid PCA will be started in the recovery room and stay with the patient until she or he does not rely on it any more. Usually, the patients keep the PCA for the first two postoperative days.
  The cumulative morphine milligram equivalent dose will be calculated from the Piritramid PCA. The PCA saves each application date and amount. This data will be gathered at the time, when the patient does not rely on the PCA any more. The Piritramid PCA will be only used in-house.
Rescue medication | The Piritramid-PCA is provided as long as requested by the patient during his in-house stay. We expect the patient to request rescue medication within the first 24 hours after surgery
  Time to first rescue medication. Rescue medication is defined as the first Piritramid application through the PCA system by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian F Baumbach, MD, Principal Investigator — Ludwig-Maximilians - University of Munich

IPD SHARING:
Plan to Share IPD: Undecided
If requested for a reasonable reason yes